CLINICAL TRIAL: NCT06074978
Title: Radiological Early Detection of Lung Cancer In Patients With Chronic Chest Diseases.
Brief Title: Early Detection of Lung Cancer In Patients With Chronic Chest Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hend Mohamed Sayed Mohamed, Lecture of chest diseases, Assiut University
Other Study IDs: LDCT &chest diseases
Record Dates: First submitted 2023-10-01; First posted 2023-10-10 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Chest--Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* To evaluate the effectiveness of LDCT in detecting early-stage lung cancer in patients with chronic lung conditions compared to standard chest x-rays.
* To improve lung cancer outcomes through optimized use of radiological technologies for early detection in high-risk patients with pre-existing lung conditions.

DETAILED DESCRIPTION:
The early detection of lung cancer is crucial, as it is one of the most common and deadly types of cancer worldwide. Early detection is especially important in patients with chronic chest diseases, as these underlying conditions can make lung cancer more difficult to diagnose at later stages. Radiological imaging techniques play a key role in the early detection of lung cancer in this high-risk patient population.

Recent advances in imaging technologies have improved our ability to detect small lung abnormalities indicative of cancer at earlier stages, even before symptoms appear . Techniques such as low-dose CT scanning have been shown to reduce lung cancer mortality by up to 20% compared to chest radiography alone . Advanced imaging allows clinicians to identify subtle nodules or masses in the lungs that may represent cancer .

Determining the type, size, and extent of lung lesions is important for prognosis and treatment planning . Imaging technologies help characterize lesions as benign or malignant and determine cancer stage . This information guides decisions around surgery, chemotherapy, radiation therapy, or other interventions .

Early detection through radiological screening has been associated with improved survival rates for lung cancer patients with chronic lung diseases . Screening finds a higher portion of early-stage, potentially curable cancers in this high-risk group . Overall, advanced imaging techniques play a vital role in the early detection and management of lung cancer in patients with underlying chronic chest conditions.

ELIGIBILITY:
Inclusion Criteria:

1- Chronic chest diseases Patients .

Exclusion Criteria:

1 - Age: less than 45 years. 2-Patients diagnosed with lung cancer 3-Unstable patients or need for ICU admission

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: After taking the informed consent, full history was taken from all patients participating in the study. Detailed clinical examination and routine laboratory investigations (complete blood count, liver function test, urea, creatinine and ESR) will be done.
  * Radiological imaging technologies -Low Dose Computed tomography (CT scans), chest x-rays These are used to detect and characterize lung abnormalities.
  * Pulmonary function tests - Spirometry volume measurements, diffusion capacity testing. These assess lung health and function in patients with chronic lung conditions
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Detection early-stage lung cancer (Stage I/II) • Lung • Lung cancer mortality rate | baseline
  By LDCT

SECONDARY OUTCOMES:
• Diagnostic accuracy of imaging modalities • Positive predictive value of screening tests • Rate of unnecessary invasive procedures • Identification of high-risk subgroups | baseline
  BY statiscal anylasis from results

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa sayed, lecture, Study Chair — Assiut University

REFERENCES:
- [Background] Balkan A, Bulut Y, Fuhrman CR, Fisher SN, Wilson DO, Weissfeld JL, Sciurba FC. COPD phenotypes in a lung cancer screening population. Clin Respir J. 2016 Jan;10(1):48-53. doi: 10.1111/crj.12180. Epub 2014 Jul 28. PMID 24989058
- [Background] Jogi J, Markstad H, Tufvesson E, Bjermer L, Bajc M. The added value of hybrid ventilation/perfusion SPECT/CT in patients with stable COPD or apparently healthy smokers. Cancer-suspected CT findings in the lungs are common when hybrid imaging is used. Int J Chron Obstruct Pulmon Dis. 2014 Dec 18;10:25-30. doi: 10.2147/COPD.S73423. eCollection 2015. PMID 25565797